CLINICAL TRIAL: NCT02466542
Title: Analgesic Effect of Intraoperative Esmolol in Mastectomies: Single Center, Prospective, Double-blind, Randomized and Placebo Controlled Study
Brief Title: Analgesic Effect of Intraoperative Esmolol in Mastectomies
Acronym: Esmobreast
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, MD, TSA, Hospital de Base
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HBase
Record Dates: First submitted 2015-06-05; First posted 2015-06-09 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Postoperative Pain
Keywords: Esmolol; Pain; Anesthesia; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia | interventions — Sodium Chloride; esmolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Placebo Comparator): Patients in placebo group will receive general balanced inhaled anesthesia with sevoflurane and remifentanil and a saline 0,9% infusion pump.
  Interventions: Drug: Placebo group
- Esmolol group (Active Comparator): Patients in esmolol group will receive general balanced inhaled anesthesia with sevoflurane and remifentanil and a bolus infection of esmolol 500 mgc/kg followed by a continuous infusion of esmolol 100 mcg/kg/min
  Interventions: Drug: Esmolol group

INTERVENTIONS:
Drug: Placebo group — Patients will receive regular general anesthesia
  Other Names: Saline
  Arms: Placebo group
Drug: Esmolol group — Patients will receive regular general anesthesia plus esmolol infusion
  Other Names: Esmolol
  Arms: Esmolol group

SUMMARY:
This study aims to compare the quality of perioperative analgesia of esmolol in patients undergoing mastectomy.

DETAILED DESCRIPTION:
Controlled hypotension is an anesthetic-surgical approach that matches the reversible and deliberate reduction in blood pressure during surgery period which aims to achieve values below 50% of normal values or mean arterial pressure (MAP) from 50 to 65 mmHg.

This technique is especially beneficial in patients undergoing procedures requiring control of bleeding for proper surgical field. The method provides a better view of anatomical structures, reduced surgical time and a significant decrease in the need for blood transfusions, with the added benefit of preventing possible complications from it.

Several drugs have been used in this scenario, as halogenated, opioids, alpha-2-agonists and beta-blockers, among which the esmolol emerges as effective and promising drug.

Esmolol is a selective beta-blocker whose action inhibits preferably the beta type 1 receptors with decreased heart rate (HR) and cardiac inotropic and consequent decrease in consumption of myocardial oxygen. Its half-life of distribution is approximately 2 minutes, the elimination half-life of 9 minutes with 55% protein bound. The duration is short due to rapid metabolism by hydrolysis by esterases in plasma and results in an inactive metabolite with negligible amounts of methanol. It has low solubility, which limits their passage through the blood-brain and placental barrier. Thanks to these features, the esmolol constitutes the most appropriate beta-blocker for intravenous use under continuous infusion.

The use of a selective beta-blocking agent continuously infused intraoperative period as well as promoting adequate blood pressure control in the controlled hypotension, it has additional advantages over other anesthetic agents, such as cardioprotection obtained by suppressing the cardiovascular response to catecholamines released during stress surgical and sympathetic stimulation resulting from laryngoscopy and tracheal intubation. The suppression of cardiovascular adrenergic response allows better coronary perfusion with proven benefits in reducing the incidence of perioperative myocardial ischemia and influence on mortality and morbidity of patients, especially coronary and high risk for ischemic phenomena. There are also several studies that demonstrate the importance of esmolol in the control and prevention of sympathetic response during extubation, better hemodynamics during induction, maintenance and emergence from anesthesia, fewer complications, lower incidence of perioperative nausea, time decreased from room to stay anesthetic recovery and, due to reduced cardiac work, action prolongation of neuromuscular blockers and opioids, saving their use. There are still ongoing studies with important indications that there is potentiation of analgesia and the hypnotic component of anesthesia with the use of esmolol.

Opioid analgesics are commonly used in clinical practice for the treatment of perioperative pain. However, many side effects are associated with its use, such as respiratory depression, nausea, vomiting, drowsiness, itching, urinary retention, constipation, hyperalgesia and impaired immune function. Therefore, alternative techniques and drugs have been used to replace their use. In recent years, the use of adjuvant drugs is becoming more popular in perioperative medicine and anesthesia, as NMDA inhibitors, local anesthetics intravenous, agonists alpha2 and beta-blockers. Some authors is likely pointing analgesic effect of intraoperative infusion of esmolol.

In this context, esmolol emerges as a drug insurance and significant effects, with impact on the quality of the anesthetic technique and the use of which should be further studied and expanded.

The patients underwent a prospective, randomized, double blind, and placebo controlled study in which the examiners responsible for intra and post-operative will not know which group they were randomly allocated: C group (n = 30) and E group (n = 30).

Both groups will receive general inhaled balanced anesthesia with sevoflurane and remifentanil.

Rapid infusion of 0.9% saline 500 ml, in both groups. In the E group is added to this solution the loading dose of esmolol with 500 mcg/kg and in group C will only be infused saline 0.9% . One infusion pump containing the result of randomization: Esmolol 100 mcg/kg/min (E group) and saline (C group).

In the clinical record, the following information will be emphasized: Blood pressure and heart rate intraoperative, perioperative side effects, quantify pain by Visual Analogue Scale (VAS) (ranging from 0 to 10 cm, zero being found when the patient is no pain and ten, with maximum or unbearable pain), Verbal Rating Scale (VRS), consisting of a list of phrases (no pain, mild pain, moderate pain, intense pain, maximum pain) and qualification of pain assessed by the amount of analgesics required postoperatively and the time to request them.

The results were analyzed statistically with the Statistical Package for Social Sciences (SPSS) version 22 (SPSS Inc., Chicago, IL, EUA) using parametric and nonparametric tests, depending on the nature of the variables studied. Data were tested for normality using the Shapiro-Wilk test. Measures of central tendency (means) and dispersion (standard deviation) were used. The level of significance was set at < 0.05. The following tests were used: Mann-Whitney test for age, duration of anesthesia and surgery, time to first analgesic supplementation, total amount of analgesics, pain intensity; Student t-test for weight and height.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, aged 18 to 75 years, electively scheduled to perform mastectomy in the Base Hospital of the Federal District;
* Physical State 1 or 2 the American Society of Anesthesiology (ASA);

Exclusion Criteria:

* Patients under the age of 18 years and above 75 years;
* Patients with unstable angina
* Patient with poorly controlled asthma
* Substance abuse
* Sinus bradycardia
* Heart failure, greater than first degree atrioventricular block
* Pregnant women
* Patients with allergy to dipyrone, morphine;
* Patients with chronic pain;
* Patients with severe hepatic disease;
* Patients with severe kidney disease;
* Patients with neurological diseases;
* Included patients in other clinical studies currently or in the past three months under general anesthesia;
* Patients who refuse to participate in the study;
* Any other condition that, in the opinion of the investigator, may pose a risk to the patient or interfere with the study objectives;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analogue Scale | Within the first 24 hours after surgery
  Quantify pain by Visual Analogue Scale (VAS, ranging from 0 to 10 cm, zero being found when the patient is no pain and ten, with maximum or un bearable pain

SECONDARY OUTCOMES:
Pain Scores on the Verbal Rating Scale | Within the first 24 hours after surgery
  Verbal Rating Scale (VRS), consisting of a list of phrases (no pain, mild pain, moderate pain, intense pain, maximum pain)
Analgesics consumption in post-operative | Within the first 24 hours after surgery
  Qualification of pain assessed by the amount of analgesics required postoperatively and the time to request them
Analgesic consumption during surgery | During the surgery
  The amount of intravenous and inhaled anesthetics consumed during surgery
Number of participants with adverse events as a measure of safety and tolerability | During the surgery
  Intraoperative hemodynamic stability analysis through the incidence of tachycardia, hypertension, bradycardia, hypotension and consumed vasopressors
Number of participants with adverse events as a measure of safety and tolerability | Within the first 24 hours after surgery
  Incidence of adverse effects such as time of awakening, nausea, vomiting, pruritus, urinary retention, drowsiness

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio T Mendonca, MD, TSA, Principal Investigator — Hospital de Base do Distrito Federal
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Celebi N, Cizmeci EA, Canbay O. [Intraoperative esmolol infusion reduces postoperative analgesic consumption and anaesthetic use during septorhinoplasty: a randomized trial]. Rev Bras Anestesiol. 2014 Sep-Oct;64(5):343-9. doi: 10.1016/j.bjan.2013.10.013. Epub 2014 Jun 21. Portuguese. PMID 25168439
- [Background] Kim Y, Hwang W, Cho ML, Her YM, Ahn S, Lee J. The effects of intraoperative esmolol administration on perioperative inflammatory responses in patients undergoing laparoscopic gastrectomy: a dose-response study. Surg Innov. 2015 Apr;22(2):177-82. doi: 10.1177/1553350614532534. Epub 2014 May 6. PMID 24803523
- [Derived] Mendonca FT, Volpe Junior JF, Tramontini AJ, DE Carvalho LS, Sposito AC. Intraoperative infusion of esmolol reduces the incidence and intensity of post-mastectomy pain syndrome. Minerva Anestesiol. 2022 May;88(5):414-415. doi: 10.23736/S0375-9393.21.16152-8. Epub 2021 Oct 12. No abstract available. PMID 34636226
- [Derived] Mendonca FT, Tramontini AJ, Miake HI, Seixas LF, de Carvalho LSF, Sposito AC. Intra-operative esmolol and pain following mastectomy: A randomised clinical trial. Eur J Anaesthesiol. 2021 Jul 1;38(7):735-743. doi: 10.1097/EJA.0000000000001512. PMID 33831899